CLINICAL TRIAL: NCT02068690
Title: Safety, Tolerability, and Pharmacokinetics of Single Rising Oral Doses of BI 425809 in Healthy Male Subjects (Partially Randomised, Single-blind, Placebo-controlled) and Investigation of Relative Bioavailability and Food Effect of BI 425809 (Open-label, Randomised, Three-way Crossover)
Brief Title: Safety, Tolerability, and Pharmacokinetics of Single Doses BI 425809
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 1346.1; 2013-004937-34 (EudraCT Number: EudraCT)
Record Dates: First submitted 2014-02-20; First posted 2014-02-21 (Estimated); Last update posted 2024-09-20 (Actual); Status verified 2024-09

CONDITIONS: Healthy
MeSH Terms: interventions — BI 425809

ARMS (2):
- BI 425809 single rising dose (Experimental): BI 425809 powder for oral solution (PfOS) in single rising doses
  Interventions: Drug: BI 425809 PfOS; Drug: Placebo
- BI 425809 Crossover (Experimental): Bioavailability of BI 425809 PfOS
  Interventions: Drug: Placebo; Drug: BI 425809 tablet; Drug: BI 425809 PfOS

INTERVENTIONS:
Drug: BI 425809 PfOS — BI 425809 PfOS
  Other Names: Iclepertin
  Arms: BI 425809 single rising dose
Drug: Placebo — Placebo
  Arms: BI 425809 single rising dose
Drug: Placebo — Placebo
  Arms: BI 425809 Crossover
Drug: BI 425809 tablet — BI 425809 tablet
  Other Names: Iclepertin
  Arms: BI 425809 Crossover
Drug: BI 425809 PfOS — BI 425809 PfOS
  Other Names: Iclepertin
  Arms: BI 425809 Crossover

SUMMARY:
To investigate safety, tolerability, and pharmacokinetics of BI 425809 following single rising doses of BI 425809 in healthy male volunteers; To explore dose proportionality of BI 425809 as oral drinking solution; To investigate relative bioavailability of BI 425809 oral drinking solution fasted compared to BI 425809 tablet fasted and tablet fed

ELIGIBILITY:
Inclusion criteria:

* Healthy male subjects
* Age 18 to 45 years (incl.)
* Body mass index (BMI) 18.5 to 29.9 kg/m2 (incl.)
* Subject must be able to understand and comply with study requirements

Exclusion criteria:

* Any finding in the medical examination (including blood pressure (BP), pulse rate (PR) or electrocardiogram (ECG)) deviating from normal and judged clinically relevant by the investigator
* Repeated measurement of systolic blood pressure <90 or >140 mmHg, or diastolic blood pressure <50 or >90 mmHg, or pulse rate <50 or >90
* Any laboratory value outside the reference range that the investigator considers to be of clinical relevance
* Any evidence of a concomitant disease judged clinically relevant by the investigator
* Gastrointestinal, hepatic, renal, respiratory, cardiovascular, metabolic, immunological or hormonal disorders
* Surgery of the gastrointestinal tract that could interfere with kinetics of the study drug(s)
* Diseases of the central nervous system (such as epilepsy), other neurological disorders or psychiatric disorders

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 83 (Actual)
Dates: Start 2014-03; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
frequency [N(%)] of subjects with drug related adverse events (AEs) | up to 18 days

SECONDARY OUTCOMES:
Cmax (maximum measured concentration of the analyte in plasma) | up to 192 hours
AUC0-infinity (area under the concentration-time curve of the analyte in plasma over the time interval from 0 extrapolated to infinity) | up to 192 hours

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (1):
- 1346.1.1 Boehringer Ingelheim Investigational Site, Ingelheim, Germany

REFERENCES:
- [Derived] Moschetti V, Desch M, Goetz S, Liesenfeld KH, Rosenbrock H, Kammerer KP, Wunderlich G, Wind S. Safety, Tolerability and Pharmacokinetics of Oral BI 425809, a Glycine Transporter 1 Inhibitor, in Healthy Male Volunteers: A Partially Randomised, Single-Blind, Placebo-Controlled, First-in-Human Study. Eur J Drug Metab Pharmacokinet. 2018 Apr;43(2):239-249. doi: 10.1007/s13318-017-0440-z. PMID 29076028